CLINICAL TRIAL: NCT06485128
Title: Investigating Multimodally Endothelial Dysfunction in Ocular and Systemic Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: S63649
Record Dates: First submitted 2023-10-05; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2023-09

CONDITIONS: Kidney Diseases; Diastolic Heart Failure; Small Vessel Disease; Glaucoma
MeSH Terms: conditions — Kidney Diseases; Heart Failure, Diastolic; Glaucoma | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Chronic kidney disease (Other)
  Interventions: Diagnostic Test: Optical coherence tomography(-angiography) OCT(A); Diagnostic Test: Fundus pictures; Diagnostic Test: DVA 3.0; Diagnostic Test: Hyperspectral retinal images; Diagnostic Test: SphygmoCor; Diagnostic Test: Sphygmomanometer; Diagnostic Test: Blood sample; Diagnostic Test: Skin biopsy; Diagnostic Test: Neuropsychological examination
- Diastolic heart failure (Other)
  Interventions: Diagnostic Test: Optical coherence tomography(-angiography) OCT(A); Diagnostic Test: Fundus pictures; Diagnostic Test: DVA 3.0; Diagnostic Test: Hyperspectral retinal images; Diagnostic Test: SphygmoCor; Diagnostic Test: Sphygmomanometer; Diagnostic Test: Blood sample; Diagnostic Test: Skin biopsy; Diagnostic Test: Neuropsychological examination
- Neuronal small vessel disease (Other)
  Interventions: Diagnostic Test: Optical coherence tomography(-angiography) OCT(A); Diagnostic Test: Fundus pictures; Diagnostic Test: DVA 3.0; Diagnostic Test: Hyperspectral retinal images; Diagnostic Test: SphygmoCor; Diagnostic Test: Sphygmomanometer; Diagnostic Test: Blood sample; Diagnostic Test: Skin biopsy; Diagnostic Test: Neuropsychological examination
- Glaucoma (Other)
  Interventions: Diagnostic Test: Optical coherence tomography(-angiography) OCT(A); Diagnostic Test: Fundus pictures; Diagnostic Test: DVA 3.0; Diagnostic Test: Hyperspectral retinal images; Diagnostic Test: SphygmoCor; Diagnostic Test: Sphygmomanometer; Diagnostic Test: Blood sample; Diagnostic Test: Skin biopsy; Diagnostic Test: Neuropsychological examination
- Healthy patients (Other)
  Interventions: Diagnostic Test: Optical coherence tomography(-angiography) OCT(A); Diagnostic Test: Fundus pictures; Diagnostic Test: DVA 3.0; Diagnostic Test: Hyperspectral retinal images; Diagnostic Test: SphygmoCor; Diagnostic Test: Sphygmomanometer; Diagnostic Test: Blood sample; Diagnostic Test: Skin biopsy; Diagnostic Test: Neuropsychological examination

INTERVENTIONS:
Diagnostic Test: Optical coherence tomography(-angiography) OCT(A) — OCTA is a non-invasive diagnostic tool capable of generating cross-sectional coupes of the retina and choroid. Novel algorithms allow to render a 3-dimensional model of the ocular microcirculation based merely on the motion contrast of the circulating blood.
Diagnostic Test: Fundus pictures — Visucam (Zeiss), Topcon NW8 fundus camera, NFC 600 (Crystalvue)
Diagnostic Test: DVA 3.0 — IMEDOS GmbH
Diagnostic Test: Hyperspectral retinal images — Ximea SNm4x4 hyperspectral snapshot camera
Diagnostic Test: SphygmoCor — Sphygmocor Excell
Diagnostic Test: Sphygmomanometer — For the measurement of the blood pressure.
Diagnostic Test: Blood sample — For both routine cardiovascular health biomarkers as well as genetic markers (DNA, mRNA, miRNA).
Diagnostic Test: Skin biopsy — Spatial proteomics and transcriptomics for endothelial function.
Diagnostic Test: Neuropsychological examination — Moca, Stroop color word test, concept shifting test, COWAT, (R)AVLT, Beck depression inventory, GDS

SUMMARY:
To explore the distribution of retinal vasculature parameters in patients with different subtypes of cardiovascular and ocular disease.

DETAILED DESCRIPTION:
In this interventional cohort study, the investigators aim to evaluate retinal vascular function as assessed by optical coherence tomography angiography, fundus photography and dynamic vessel analysis in patients who share microvascular involvement of their pathology (e.g. chronic kidney disease, cardiac decompensation, neuronal small vessel disease and glaucoma) and age-matched healthy controls. Plasm and skin samples for comparative proteomics and transcriptomics are also taken.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with a confirmed or suspect diagnosis of glaucoma based on intra-ocular eye pressure, visual field defect and structural optic nerve changes, regardless their age.
* Adult patients with chronic kidney disease regardless their age.
* Adult patients with heart failure with preserved ejection fraction (HFpEF), regardless their age: symptomatic heart failure with Left Ventricle Ejection Fraction > 50% AND BNP > 35 pg/ml (or NT-proBNP>125 pg/ml) OR signs of diastolic dysfunction according to the European Society of Cardiology guidelines 2016
* Adult patients with confirmed small vessel disease as is diagnosed on routine neurological imaging, regardless their age.
* People without history or track record of any relevant pathology, including cardiovascular and renal diseases, regardless their age
* Capable and willing to participate (informed consent)

Exclusion Criteria:

* Diabetes
* Personal medical history of retinal neovascularization.
* Unable or unwilling to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2021-07-06 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Relative distribution of retinal endothelial reactivity, flow index, vessel density in the different subpopulations. | 3 years

SECONDARY OUTCOMES:
Diagnostic performance of the aforementioned parameters to distinguish the different subpopulations. | 3 years
The association between these parameters and (1) the presence of risk factors for cardiovascular disease (including biomarkers) and (2) risk factors for disease progression and (3) neuropsychological functioning | 3 years
Physiological behaviour of retinal vasculature under cardiovascular stress. | 3 years
Histopathological correlates in dermal microvasculature | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Ingeborg Stalmans, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- Universitaire Ziekenhuizen UZ/KU Leuven, Leuven, Vlaams-Brabant, Belgium